CLINICAL TRIAL: NCT05853211
Title: Therapeutic Effects of Class II Elastics on Aligners in Different Vertical Skeletal Patterns in Adult Patients: Retrospective Study.
Brief Title: Therapeutic Effects of Class II Elastics on Aligners in Different Vertical Skeletal Patterns
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, VANDE VANNET Bart, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023PI022
Record Dates: First submitted 2023-04-13; First posted 2023-05-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Malocclusion, Angle Class II
Keywords: aligner; inter-arch elastic; orthodontic; class II malocclusion; adult; clear aligner; orthodontic appliance; Invisalign; class II elastics; angle class II malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clear aligner: Patient with class II malocclusion, treated with class II elastics on aligners
  Interventions: Combination Product: Aligner and inter-arch elastics
- Fixed appliance: Patient with class II malocclusion, treated with class II elastics on fixed appliance

INTERVENTIONS:
Combination Product: Aligner and inter-arch elastics — Correction of class II malocclusion by class II elastics on clear aligners
  Groups: Clear aligner

SUMMARY:
The objective is to compare the dento-alveolar therapeutic effects of wearing class II inter-arch traction elastics on aligners versus multi-brackets in an adult population. The principal hypothesis is no significant difference in therapeutic effects of using inter-arch elastics on aligners versus multi-brackets.

DETAILED DESCRIPTION:
It is a non-interventional research involving the human person, research on existing data and / samples in the field of dentofacial orthopedics. This study analyzes the effects of rubber bands when combined with aligners in adult patients. This is a comparative retrospective study of radiographs and casts before and after orthodontic treatment. The patients studied are in Angle class II and adults. Two groups are analysed: patients treated with fixed (vestibular multi-attachment) and removable (Invisalign-type aligners) appliances.

ELIGIBILITY:
Inclusion Criteria:

* CVM stage 5 on lateral teleradiography (end of growth)
* Angle Class II
* Treatments with rubber bands for inter-arch traction
* End of treatment in class I

Exclusion Criteria:

* Incomplete data
* Treatment with extractions, mini-screws, mini-plate or ortho-surgical treatment
* Dental agenesis (excluding wisdom teeth)
* Cranial-facial syndromes

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult with class II malocclusion treated with class II elastics
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in IMPA Mandibular incisor angle (degrees) | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months.
  Angle between the mandibular plane and the lower incisor axis: position of the lower incisor in relation to the mandible

SECONDARY OUTCOMES:
Sex | 1 month
  Sex
Duration of treatment | 24 months
  Treatment time duration in month
Change in interproximal dental size | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Interproximal size in mm
Change in skeletal sagittal pattern ANB angle | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : angle between A, Na (nasion) and B in degrees
Change in skeletal sagittal pattern Ao-Bo | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : mesure in mm between Ao and Bo
Change in skeletal vertical pattern : FMA | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : angle in degrees between franckfort plan and mandibular plan.
Change in skeletal vertical pattern : Sn Gogn | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : angle in degrees between SN and GoGn
Change in faciale anterior height | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements of faciale anterior height
Change in faciale posterior height | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements of faciale posterior height
Change in index Faciale height | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements, index HFP (faciale posterior heigth)/ HFA (faciale anterior height)
Change in nterincisal angle | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : measurement between manxillary and mandibular incisors.
Change in plan of occlusion | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Cephalometric measurements : angle between SN and Op
Age at the beginning of treatment | 1 month
  Age
Age at the end of treatment | 24 months
  Age
Change in von Spee curve | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : it is the average of the distance between the highest point of the deepest cusp and the occlusal plane.
Change in overall crowding | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : comparison of the sum of the mesiodistal diameters of 35 to 45 and the arch perimeter from the mesial face of 36 to the mesial face of 46.
Change in overjet | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : in mm
Change in overbite | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : in mm
Change in arch length | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : distance between inter incisal point and mesiale face of 6.
CHange in class II quantity | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : inter canine and inter molar relations
Change in space required | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : sum of all mesiodistal diameter.
Change in inter canine distance | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : distance between the canine in mm
Change in inter premolar distance | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : distance between the premolars
Change in inter molar distance | First : just before the beginning of treatment; Second : just after the end of orthodontic treatment. An average of 18 months
  Measurements on impressions : distance between the molars

CONTACTS AND LOCATIONS:
Overall Officials: Bart VANDE VANNET, Study Director — Central Hospital, Nancy, France
Locations (1):
- DEON, Nancy, Lorraine, France

REFERENCES:
- [Background] Janson G, Sathler R, Fernandes TM, Branco NC, Freitas MR. Correction of Class II malocclusion with Class II elastics: a systematic review. Am J Orthod Dentofacial Orthop. 2013 Mar;143(3):383-92. doi: 10.1016/j.ajodo.2012.10.015. PMID 23452973
- [Background] Robertson L, Kaur H, Fagundes NCF, Romanyk D, Major P, Flores Mir C. Effectiveness of clear aligner therapy for orthodontic treatment: A systematic review. Orthod Craniofac Res. 2020 May;23(2):133-142. doi: 10.1111/ocr.12353. Epub 2019 Nov 13. PMID 31651082
- [Background] Zheng M, Liu R, Ni Z, Yu Z. Efficiency, effectiveness and treatment stability of clear aligners: A systematic review and meta-analysis. Orthod Craniofac Res. 2017 Aug;20(3):127-133. doi: 10.1111/ocr.12177. Epub 2017 May 26. PMID 28547915
- [Background] Lombardo L, Colonna A, Carlucci A, Oliverio T, Siciliani G. Class II subdivision correction with clear aligners using intermaxilary elastics. Prog Orthod. 2018 Sep 1;19(1):32. doi: 10.1186/s40510-018-0221-5. PMID 30171391
- [Background] Dianiskova S, Rongo R, Buono R, Franchi L, Michelotti A, D'Anto V. Treatment of mild Class II malocclusion in growing patients with clear aligners versus fixed multibracket therapy: A retrospective study. Orthod Craniofac Res. 2022 Feb;25(1):96-102. doi: 10.1111/ocr.12500. Epub 2021 May 31. PMID 34013659
- [Background] Duncan LO, Piedade L, Lekic M, Cunha RS, Wiltshire WA. Changes in mandibular incisor position and arch form resulting from Invisalign correction of the crowded dentition treated nonextraction. Angle Orthod. 2016 Jul;86(4):577-83. doi: 10.2319/042415-280.1. Epub 2015 Dec 4. PMID 26636248
- [Background] Amm E, El Amm C, Vaden J. Effect of Class II elastics on different mandibular arch preparation stabilized with aligners and stainless-steel wires: A FEM study. Orthod Craniofac Res. 2022 Nov;25(4):520-529. doi: 10.1111/ocr.12564. Epub 2022 Jan 27. PMID 35015923
- [Background] Rongo R, Dianiskova S, Spiezia A, Bucci R, Michelotti A, D'Anto V. Class II Malocclusion in Adult Patients: What Are the Effects of the Intermaxillary Elastics with Clear Aligners? A Retrospective Single Center One-Group Longitudinal Study. J Clin Med. 2022 Dec 9;11(24):7333. doi: 10.3390/jcm11247333. PMID 36555949
- [Background] Deregibus A, Tallone L, Rossini G, Parrini S, Piancino M, Castroflorio T. Morphometric analysis of dental arch form changes in class II patients treated with clear aligners. J Orofac Orthop. 2020 Jul;81(4):229-238. doi: 10.1007/s00056-020-00224-8. Epub 2020 Apr 14. PMID 32291482
- [Background] Liu X, Cheng Y, Qin W, Fang S, Wang W, Ma Y, Jin Z. Effects of upper-molar distalization using clear aligners in combination with Class II elastics: a three-dimensional finite element analysis. BMC Oral Health. 2022 Dec 1;22(1):546. doi: 10.1186/s12903-022-02526-2. PMID 36456944
- [Background] Baccetti T, Franchi L, McNamara JA Jr. An improved version of the cervical vertebral maturation (CVM) method for the assessment of mandibular growth. Angle Orthod. 2002 Aug;72(4):316-23. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12169031
- [Background] Marshall SD, Caspersen M, Hardinger RR, Franciscus RG, Aquilino SA, Southard TE. Development of the curve of Spee. Am J Orthod Dentofacial Orthop. 2008 Sep;134(3):344-52. doi: 10.1016/j.ajodo.2006.10.037. PMID 18774080
- [Background] Fawaz P, Amm E, Khoury E. The curve of Spee and its levelling in different vertical skeletal patterns: A 3D set-up study. Int Orthod. 2021 Dec;19(4):659-668. doi: 10.1016/j.ortho.2021.08.003. Epub 2021 Aug 31. PMID 34479824
- [Background] Adel SM, Vaid NR, El-Harouni N, Kassem H, Zaher AR. Digital model superimpositions: are different software algorithms equally accurate in quantifying linear tooth movements? BMC Oral Health. 2022 Mar 31;22(1):103. doi: 10.1186/s12903-022-02129-x. PMID 35361187